CLINICAL TRIAL: NCT02797444
Title: Advance Care Planning for Critical Care - A Prelude to Breaking Barriers
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 106476
Record Dates: First submitted 2016-03-31; First posted 2016-06-13 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2016-02

CONDITIONS: Advance Care Planning; End of Life Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: semi-structured interviews

SUMMARY:
Advance Care Planning (ACP) is a process of 'reflection and communication, in which a person with decision-making capacity makes decisions regarding their future health and/or personal care in the event that they become incapable of consenting to or refusing treatment' Most Canadians have not planned for end-of-life Care and are at risk of aggressive medical care that may not be compatible with their wishes. This study aims to systematically evaluate local barriers to making personal choices with regards to life support interventions that can be provided in the contemporary Intensive Care Unit.

DETAILED DESCRIPTION:
HYPOTHESIS: The overarching hypothesis is that the average layperson lacks sufficient knowledge about the aggressive life support measures used routinely in contemporary Critical Care to make informed decisions for themselves and their loved ones. Considering that most Canadians have not even heard of the term Advance Care Planning, it is likely that there is a gap in their knowledge and expectations of Critical Care. Such a gap can be bridged through education - the only caveat being that the individual should be in full possession of their faculties and can make informed decisions. This point is critical.

Thus this study uses a mixed methods (qualitative and quantitative) research design to address the following questions: 1) What is the state of knowledge about Critical Care interventions among healthy elderly laypersons in London, Ontario? 2) What are the barriers to formulating ACPs? 3) What opportunities exist for increasing ACP in the healthy elderly population? The primary objective of this proposal is to assess public knowledge of Critical Care interventions (and their outcomes) from the perspective of making Advance Care Plans. Secondary Objectives are 1) To evaluate local barriers to Advance Care Planning 2) To determine effective modes of education for Advance Care Planning that could be used for the community and in our hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Members from the community who are i) > 55 yrs of age, ii) living in London Middlesex community, iii) not housebound, iv) in apparent good health and iv) have the ability to make independent decisions for themselves

Exclusion Criteria:

* Factors that preclude a meaningful interview (such as cognitive impairment, aphasia, profound hearing impairment, language barriers) or anticipated emotional burden with the proposed topic.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy lay persons living at home in London, ON.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Lay person perception and knowledge of various Critical Care interventions | 1 year
  This is a qualitative study. The primary objective of this proposal is to assess public knowledge of Critical Care interventions (and their outcomes) from the perspective of making Advance Care Plans. Examples of such interventions include but are not limited to Cardiopulmonary resuscitation, mechanical ventilation, dialysis and artificial feeding. Outcomes involve lay person knowledge, beliefs and perceptions of Critical care from the perspective of making Advance Care Plans.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Taneja, MBBS, Principal Investigator — London Health Sciences Centre
Locations (2):
- Canada (2):
  - Dr. Ravi Taneja, London, Ontario
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teixeira AA, Hanvey L, Tayler C, Barwich D, Baxter S, Heyland DK; Canadian Researchers at End of Life Network (CARENET). What do Canadians think of advanced care planning? Findings from an online opinion poll. BMJ Support Palliat Care. 2015 Mar;5(1):40-7. doi: 10.1136/bmjspcare-2013-000473. Epub 2013 Oct 4. PMID 24644188
- [Derived] Taneja R, Faden LY, Schulz V, Rawal A, Miller K, Bishop KA, Lingard L. Advance care planning in community dwellers: A constructivist grounded theory study of values, preferences and conflicts. Palliat Med. 2019 Jan;33(1):66-73. doi: 10.1177/0269216318803487. Epub 2018 Oct 4. No abstract available. PMID 30284950